CLINICAL TRIAL: NCT00335088
Title: Local Moxifloxacin and Povidone Iodine Versus Povidone Iodine Alone as a Prophylaxis Before Eye Operations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4780506
Record Dates: First submitted 2006-06-05; First posted 2006-06-08 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-03

CONDITIONS: Eye Infections
Keywords: Prophylaxis,; Intraocular surgery; Lacrimal sac; Eye lid; No conditions
MeSH Terms: conditions — Eye Infections | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Moxifloxacin and Povidone Iodine vs Povidone Iodine

SUMMARY:
The hypothesis is that povidone iodine alone is sufficient for sterilization of the lacrimal sac and eye lids before intraocular surgeries. Patients admitted for various intraocular surgeries will be randomly allocated to prophylactic local therapy with either moxifloxacin and povidone iodine or povidone iodine alone before surgery. Lacrimal sac and eye lid cultures will be obtained before the local therapy and just before surgery.

DETAILED DESCRIPTION:
Over all 500 patients admitted for various intraocular surgeries will be included in the study. The study will be prospective, double blind, placebo controlled, and randomized. Patients will be randomly allocated to prophylactic local therapy with either moxifloxacin and povidone iodine or povidone iodine alone before surgery. For patients treated with povidone iodine alone a placebo will also be given. Lacrimal sac and eye lid cultures will be obtained before the local therapy and just before surgery. All patients will be followed for 6 weeks for symptoms and signs of infection. Bacterial and fungal culture results will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years.
* Various intraocular surgeries

Exclusion Criteria:

* Need for emergency therapy, immunosuppression, any malignancy, psychomotor retardation, drug and alcohol abuse.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-06; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Type and amount of bacterial growth
Post surgery infections

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miron, MD, Study Director — HaEmek Medicak Center, Afula, Israel; Orky Halachmi, MD, Principal Investigator — HaEmek Medical Center, Afula, Israel
Locations (1):
- Ophthalmology Department, HaEmek Medical Center, Afula, Israel, Afula, Israel